CLINICAL TRIAL: NCT05947760
Title: Magnesium as an Adjuvant Agent for Postoperative Pain Control Following Periacetabular Osteotomy
Brief Title: Magnesium as an Adjuvant Agent for Postoperative Pain
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Robert Wetzel, MD, Orthopedic Trauma Surgeon, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY20230720
Record Dates: First submitted 2023-07-05; First posted 2023-07-17 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-03

CONDITIONS: Pain, Postoperative
Keywords: periacetabular osteotomy; IV magnesium sulfate; Decreased opioid usage
MeSH Terms: conditions — Pain, Postoperative | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV Magnesium Sulfate adjuvant group (Experimental): Participants in this group will receive standard-of-care procedures intraoperatively and postoperatively along with IV magnesium sulfate for pain control.
  Interventions: Drug: IV Magnesium Sulfate
- Control group (No Intervention): Participants in this group will receive standard-of-care procedures intraoperatively and post-operatively for pain control.

INTERVENTIONS:
Drug: IV Magnesium Sulfate — Participants will receive IV Magnesium Sulfate intraoperatively.
  Arms: IV Magnesium Sulfate adjuvant group

SUMMARY:
Participants are being asked to participate in this research study because they have elected to undergo periacetabular osteotomy (PAO). This research study is looking at if using IV magnesium during surgery can help to reduce pain after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing periacetabular osteotomy with or without adjuvant hip arthroscopy

Exclusion Criteria:

* illiterate or non-English speaking patients
* patients with 2nd or 3rd degree AV block
* patients with severe renal insufficiency
* patients with heart failure
* patients with bradycardia

Ages: 14 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain as measured by the Visual Analog Scale (VAS) | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, 1 year
  The VAS is a scale from 0-10 with 0 being no pain and 10 being the worst pain ever
Change in number of narcotic medications consumed as measured by the medical record review | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, 1 year

SECONDARY OUTCOMES:
Change in PROMIS scores | 2 weeks, 6 weeks, 3 months, 6 months, 1 year
  The PROMIS is a 14 item questionnaire is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. Scores are typically between 20-80, but may be 0-100.
Change in modified Harris Hip Scores (mHHS) | 2 weeks, 6 weeks, 3 months, 6 months, 1 year
  The mHHS is a scoring system for functional outcomes post periactabular osteotomies that has a scale of 0-100, 0 being the lowest functional outcome and 100 being the highest

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wetzel, MD, Principal Investigator — University Hospitals
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No